CLINICAL TRIAL: NCT03847506
Title: A Randomized, Double-blind, Multi-center Clinical Trial to Evaluate Efficacy and Safety of Ezetimibe/Rosuvastatin Combination Tablets and Candesartan Cilexetil/Amlodipine Besylate Combination Tablets
Brief Title: Evaluate Efficacy and Safety of Ezetimibe/Rosuvastatin and Candesartan Cilexetil/Amlodipine Besylate Combination Tablets
Acronym: REVERT-K
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CJ_RVZ_401
Record Dates: First submitted 2018-11-20; First posted 2019-02-20 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Hypertension, Hyperlipidemia
MeSH Terms: conditions — Hypertension; Hyperlipidemias | interventions — Ezetimibe; Rosuvastatin Calcium; candesartan cilexetil; Amlodipine

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EZE/ROS+CAN/AML (Experimental): Ezetimibe/Rosuvastatin 10 mg/10 mg and Candesartan cilexetil/Amlodipine besylate 8 mg/5 mg, once a day for 6 weeks
  Interventions: Drug: Ezetimibe/Rosuvastatin
- CAN/AML (Active Comparator): Candesartan cilexetil/Amlodipine besylate 8 mg/5 mg, once a day for 6 weeks
  Interventions: Drug: Candesartan cilexetil/Amlodipine besylate
- EZE/ROS+CAN (Active Comparator): Ezetimibe/Rosuvastatin 10 mg/10 mg + Candesartan cilexetil 8 mg, once a day for 6 weeks
  Interventions: Drug: Candesartan cilexetil

INTERVENTIONS:
Drug: Ezetimibe/Rosuvastatin — Ezetimibe/Rosuvastatin 10 mg/10 mg + Candesartan cilexetil/Amlodipine besylate 8 mg/5 mg + Candesartan cilexetil 8 mg placebo
  Other Names: Ezetimibe/Rosuvastatin 10 mg/10 mg
  Arms: EZE/ROS+CAN/AML
Drug: Candesartan cilexetil/Amlodipine besylate — Candesartan cilexetil/Amlodipine besylate 8 mg/5 mg + Ezetimibe/Rosuvastatin 10 mg/10 mg placebo + Candesartan cilexetil 8 mg placebo
  Other Names: Candesartan cilexetil/Amlodipine besylate 8 mg/5 mg
  Arms: CAN/AML
Drug: Candesartan cilexetil — Ezetimibe/Rosuvastatin 10 mg/10 mg + Candesartan cilexetil 8 mg + Candesartan cilexetil/Amlodipine besylate 8 mg/5 mg placebo
  Other Names: Candesartan cilexetil 8 mg
  Arms: EZE/ROS+CAN

SUMMARY:
To evaluate the efficacy and the safety of concomitant use of Ezetimibe/Rosuvastatin combination tablets and Candesartan cilexetil/Amlodipine besylate combination tablets compared to each combination tablet alone in patients with essential hypertension (HTN) and hyperlipidemia.

DETAILED DESCRIPTION:
To improve the ease of use of high blood pressure and hyperlipidemia to improve patient compliance and reduce the risk of cardiovascular disease.

And It is recommended to identify the need to develop a combination of Candesartan cilexetil/Amlodipine besylate combination tablets , and Ezetimibe/Rosuvastatin combination tablets.

ELIGIBILITY:
[ Inclusion Criteria ]

1. Adults aged 19 to <75 years.
2. Diagnosed with essential HTN accompanied by hyperlipidemia (average siSBP ≥140 mmHg and LDL-C ≥100 mg/dL) or being treated for the condition after the diagnosis, at Visit 1 (screening).
3. Provided the signed informed consent form voluntarily after receiving explanation of the objectives, methods and effects of the study.
4. Medically sterile or agreed to use medically acceptable contraceptive method during the study.

[ Exclusion Criteria ]

* Criteria Related to HTN and Dyslipidemia

1. Severe HTN defined as average siDBP ≥110 mmHg or average siSBP ≥180 mmHg at Visit 1 (screening).
2. The difference in BPs between those measured at both arms at Visit 1 (screening) is ≥10 mmHg for siDBP or ≥20 mmHg for siSBP.
3. LDL-C >250 mg/dL or TG ≥400 mg/dL at Visit 1 (screening).
4. Diagnosed with or suspected of secondary HTN (e.g., renovascular disease, coarctation of the aorta, hyperaldosteronism, unilateral or bilateral renal artery stenosis, Cushing's syndrome, pheochromo-cytoma, polycystic kidney disease, etc.).
5. Patients with symptomatic orthostatic HTN (difference in BPs between the value measured in supine position and the value measured in standing position is ≥20 mmHg for siSBP or ≥10 mmHg for siDBP).

   * Criteria Related to Medical History
6. Diagnosis with type 1 diabetes mellitus (DM) or uncontrolled DM (patients on insulin therapy or patients with HbA1C ≥9%).
7. Patients with severe heart disease - heart failure (NYHA Classes 3 and 4), history of ischemic cardiac disease (unstable angina, myocardial infarction), peripheral vascular diseases, percutaneous transluminal angioplasty, or coronary artery bypass graft within the recent 3 months.
8. Patients with clinically significant ventricular tachycardia, atrial fibrillation, atrial flutter, or other clinically significant arrhythmia at the discretion of the investigator.
9. History of muscular toxicity while on treatment with other HMG-CoA reductase inhibitors or fibrates.
10. History of angioedema while on treatment with ACE inhibitors or ARBs.
11. History of hypersensitivity to ARBs, dihydropyridines, or HMG-CoA reductase inhibitors.
12. Patients with hypertrophic occlusive myocardiopathy, severe occlusive coronary artery disease, aortic stenosis, hemodynamically significant aortic, or mitral valve stenosis.
13. Presence of severe cerebrovascular disorders (diagnosis of stroke, cerebral infarction, or cerebral hemorrhage within the recent 6 months).
14. History or current evidence of wasting diseases, autoimmune diseases (such as rheumatoid arthritis and systemic lupus erythematosus), or connective tissue diseases.
15. Known diagnosis of moderate or malignant retinopathy (including retinal hemorrhage, visual disturbance, and retinal microaneurysm within the recent 6 months).
16. Patients with surgical or medical gastrointestinal diseases or having received surgery that could interfere with drug absorption, distribution, metabolism, and elimination and patients with active gastritis, gastrointestinal/rectal bleeding, or diagnosed with active inflammatory bowel disease within the recent 12 months.
17. History of malignancy including leukemia and lymphoma within the recent 5 years (except for localized basal cell carcinoma of the skin).
18. Patients with any inflammatory diseases requiring chronic anti-inflammatory therapy.
19. Patients who received kidney transplant or with only one kidney.
20. Presence of biliary obstruction or cholestasis.
21. Presence of hereditary conditions such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.
22. Patients with shock.

    * Criteria Related to Clinical Laboratory Tests
23. Laboratory abnormalities as follows:

    * AST or ALT >3 x upper limit of normal (ULN);
    * Serum creatinine >1.5 x ULN.
24. History of myopathy or rhabdomyolysis (e.g., serum CK ≥5 x ULN).
25. Uncontrolled abnormal thyroid function (e.g., TSH ≥1.5 x ULN).
26. Persistent abnormal serum potassium level (e.g., serum potassium level <3.5 mmol/L or >5.5 mmol/L).
27. Patients with conditions of body fluid depletion or laboratory findings indicating clinically significant electrolyte abnormality.

    * Others
28. Needs for concomitant administration of non-study antihypertensive agents or prohibited medications during the study.
29. Pregnant or lactating women.
30. History of drug or alcohol abuse within the recent 1 year.
31. Having received other investigational product within 4 weeks prior to screening.
32. Patients considered ineligible for the study at the discretion of the principal investigator (PI) or study staff.

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
Change in sitting Systolic Blood Pressure(siSBP) from baseline after 6 weeks of study treatment | week 6
  EZE/ROS + CAN/AML arm vs. EZE/ROS + CAN arm
  Change in siSBP from baseline after 6 weeks of study treatment For the siSBP at baseline and after 6 weeks of study treatment, the mean, standard deviation, median, minimum, and maximum will be provided by treatment arm. The LS-mean change in baseline-adjusted siSBP from baseline after 6 weeks of study treatment and its standard error will be provided by treatment arm. Inter-arm comparison will be conducted using the analysis of covariance (ANCOVA) with change in siSBP as response variable and baseline siSBP and treatment arm as independent variables.
Percentage change in LDL-C levels from baseline after 6 weeks of study treatment | week 6
  EZE/ROS + CAN/AML arm vs. CAN/AML arm
  Percentage change in LDL-C levels from baseline after 6 weeks of study treatment For the percentage change in LDL-C levels at baseline and after 6 weeks of study treatment, the mean, standard deviation, median, minimum, and maximum will be provided by treatment arm. The LS-mean percentage change in baseline-adjusted LDL-C levels from baseline after 6 weeks of study treatment and its standard error will be provided by treatment arm. Inter-arm comparison will be conducted using the ANCOVA with percentage change in LDL-C levels as response variable and baseline LDL-C level and treatment arm as independent variables.

SECONDARY OUTCOMES:
Change in siSBP from baseline after 3 weeks of study treatment | week 3
  EZE/ROS + CAN/AML arm vs. EZE/ROS + CAN arm
  For the siSBP at baseline and after 3 weeks of study treatment, the mean, standard deviation, median, minimum, and maximum will be provided by treatment arm. The LS-mean change in baseline-adjusted siSBP from baseline after 3 weeks of study treatment and its standard error will be provided by treatment arm. Inter-arm comparison will be conducted using the ANCOVA with change in siSBP as response variable and baseline siSBP and treatment arm as independent variables.
Percentage changes in LDL-C levels from baseline after 3 and 6 weeks of study treatment | week 3 and week 6
  EZE/ROS + CAN/AML arm vs. EZE/ROS + CAN arm
  For the LDL-C levels at baseline and after 3 and 6 weeks of study treatment, the mean, standard deviation, median, minimum, and maximum will be provided by treatment arm. The LS-mean percentage changes in baseline-adjusted LDL-C levels from baseline after 3 and 6 weeks of study treatment and their standard error will be provided by treatment arm. Inter-arm comparisons of the percentage changes in LDL-C levels at Week 3 and Week 6 will be conducted using the ANCOVA with percentage change in LDL-C levels as response variable and baseline LDL-C level and treatment arm as independent variables.
Percentage change in LDL-C levels from baseline after 3 weeks of study treatment | week 3
  EZE/ROS + CAN/AML arm vs. CAN/AML arm
  For the percentage change in LDL-C levels at baseline and after 3 weeks of study treatment, the mean, standard deviation, median, minimum, and maximum will be provided by treatment arm. The LS-mean percentage change in baseline-adjusted LDL-C levels from baseline after 3 weeks of study treatment and its standard error will be provided by treatment arm. Inter-arm comparison will be conducted using the ANCOVA with percentage change in LDL-C levels as response variable and baseline LDL-C level and treatment arm as independent variables.
Changes in siSBPs from baseline after 3 and 6 weeks of study treatment | week 3 and week 6
  EZE/ROS + CAN/AML arm vs. CAN/AML arm
  For the siSBP at baseline and after 3 and 6 weeks of study treatment, the mean, standard deviation, median, minimum, and maximum will be provided by treatment arm. The LS-mean change in baseline-adjusted siSBP from baseline after 3 and 6 weeks of study treatment and its standard error will be provided by treatment arm. Inter-arm comparison will be conducted using the ANCOVA with change in siSBP as response variable and baseline siSBP and treatment arm as independent variables.
Percentage changes in LDL-C/HDL-C and TC/HDL-C from baseline after 3 and 6 weeks of study treatment | week 3 and week 6
  EZE/ROS + CAN/AML arm vs. CAN/AML arm
  For the LDL-C/HDL-C and TC/HDL-C at baseline and for their percentage changes after 3 and 6 weeks of study treatment, the mean, standard deviation, median, minimum, and maximum were presented by treatment arm. The LS-mean percentage changes in baseline-adjusted LDL-C/HDL-C and TC/HDL-C levels from baseline after 3 and 6 weeks of study treatment and their standard errors will be provided by treatment arm. Inter-arm comparison will be conducted using the ANCOVA with percentage changes in LDL-C/HDL-C and TC/HDL-C levels as response variables and baseline LDL-C/HDL-C and TC/HDL-C levels and treatment arm as independent variables.
Changes in siDBPs from baseline after 3 and 6 weeks of study treatment | week 3 and week 6
  Co-Endpoints
  For the siDBP at baseline and after 3 and 6 weeks of study treatment, the mean, standard deviation, median, minimum, and maximum will be provided by treatment arm. The LS-mean change in baseline-adjusted siDBP from baseline after 3 and 6 weeks of study treatment and its standard error will be provided by treatment arm. Inter-arm comparison will be conducted using the ANCOVA with change in siDBP as response variable and baseline siDBP and treatment arm as independent variables.
Proportions of subjects who achieve the treatment goal based on JNC VIII Guideline from baseline after 3 and 6 weeks of study treatment | week 3 and week 6
  Co-Endpoints
  (HTN treatment goal: <140/90 mmHg [or <150/90 mmHg for patients aged ≥60 years]) The frequencies and proportions of subjects who achieve the treatment goal based on JNC VIII Guideline from baseline after 3 and 6 weeks of study treatment will be provided by treatment arm. The differences in the proportions of subjects who achieve the treatment goal after 3 and 6 weeks of study treatment between treatment arms will be analyzed using the Pearson's chi-square test or the Fisher's exact test.
Proportions of subjects who achieve the treatment goal based on NCEP ATP III Guideline from baseline after 3 and 6 weeks of study treatment | week 3 and week 6
  Co-Endpoints
  (LDL-C treatment goal - Group I: <160 mg/dL; Group II: <130 mg/dL; and Group III: <100 mg/dL) The frequencies and proportions of subjects who achieve the treatment goal based on NCEP ATP III Guideline from baseline after 3 and 6 weeks of study treatment will be provided by treatment arm. The differences in the proportions of subjects who achieve the treatment goal after 3 and 6 weeks of study treatment between treatment arms will be analyzed using the Pearson's chi-square test or the Fisher's exact test.
Percentage changes in TC, TG, HDL-C, apolipoprotein B, and CRP levels from baseline after 3 and 6 weeks of study treatment | week 3 and week 6
  Co-Endpoints
  For the TC, TG, HDL-C, apolipoprotein B, and CRP levels at baseline and after 3 and 6 weeks of study treatment, the mean, standard deviation, median, minimum, and maximum will be provided by treatment arm. The LS-mean percentage changes in baseline-adjusted TC, TG, HDL-C, apolipoprotein B, and CRP levels from baseline after 3 and 6 weeks of study treatment and their standard error will be provided by treatment arm. Inter-arm comparisons of the percentage changes at Week 3 and Week 6 will be conducted using the ANCOVA with each percentage change in TC, TG, HDL-C, apolipoprotein B, and CRP levels as response variable and relevant baseline level and treatment arm as independent variables.

OTHER OUTCOMES:
Adverse events | Baseline, week 3 and week 6
  The safety will be evaluated for all subjects who receive at least on dose of investigational product. The number of subjects who report AEs, adverse drug reactions (ADRs), serious adverse events (SAEs), two-sided 95% CIs, incidence rate, and number of events will be provided by treatment arm. The difference between treatment arms will be analyzed using the χ2 test or Fisher's exact test. The incidences and percentages of events by severity, causality, actions taken, and outcome will be provided by treatment arm.
  All AEs will be coded per SOC and PT using the MedDRA; for each coded AE, the number of subjects, incidence rate, and number of events will be provided by treatment arm. In addition, for coded AEs, the number of subjects, incidence rate, and number of events by severity, causality, actions taken, and outcome will be provided by treatment arm

CONTACTS AND LOCATIONS:
Overall Officials: In-Ho Chae, Ph.D, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Bundang Seoul National University Hospital, Gyeonggi-do, Seongnam-si, Bundang-gu, South Korea

IPD SHARING:
Plan to Share IPD: No